CLINICAL TRIAL: NCT00451763
Title: Intravitreal Bevacizumab for Idiopathic Macular Telangiectasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 165/07
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2007-03

CONDITIONS: Retina; Telangiectasis
Keywords: Fovea centralis/pathology; Fundus oculi; Retinal neovascularization; Telangiectasis/diagnosis; Tomography, optical coherence; Vitreous Body/drug effects
MeSH Terms: conditions — Telangiectasis; Retinal Neovascularization; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Intravitreal Injection of Bevacizumab (1.25 mg/0.05ml)

SUMMARY:
Idiopathic Macular Telangiectasia is characterized by incompetent and dilated retinal capillaries in the foveolar region of unknown cause for retinal telangiectasia.

In Idiopathic Macular Telangiectasia, proliferative changes occur in the deep retinal capillary network, leading to intraretinal neovascularization that, unlike in age-related macular degeneration, seems to be retinal rather than choroidal in origin. Before the hemorrhagic and fibrotic state, these vessels may lead to exudation and decrease in the visual acuity. Long-term visual prognosis in patients with this complication may be poor and treatment with laser photocoagulation is unproven. Although newly reported treatment, by photodynamic therapy for neovascular membrane associated with Idiopathic Macular Telangiectasia, may show vision and angiographic stability in a few cases, the improvement may be transient. VEGF has been implicated as the major angiogenic stimulus responsible for neovascularization in AMD, ensuing specific anti-VEGF treatment in these cases.

The purpose of the study is to evaluate intravitreal injection of bevacizumab (1.25mg/0.05ml) in the treatment of Idiopathic Macular Telangiectasia.

ELIGIBILITY:
Inclusion Criteria:

* patients with idiopathic macular telangiectasia
* patient consent

Exclusion Criteria:

* heart attack or cerebrovascular attack
* previous treatment for others retinopathy
* media opacities that preclude visualization of the fundus
* inability to understands the implications of the protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity
Optical coherence tomography
Fluorescein angiography

CONTACTS AND LOCATIONS:
Overall Officials: Walter Y Takahashi, M.D., Study Director — University of Sao Paulo; Otacilio O Maia Jr, M.D., Principal Investigator — Sao Rafael Hospital, Monte Tabor Foudation
Locations (1):
- From the Retina and Vitreous Service, Department of Ophthalmology. Sao Rafael Hospital, Monte Tabor Foudation, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Maia OO Jr, Bonanomi MT, Takahashi WY, Nascimento VP, Takahashi BS. Intravitreal bevacizumab for foveal detachment in idiopathic perifoveal telangiectasia. Am J Ophthalmol. 2007 Aug;144(2):296-9. doi: 10.1016/j.ajo.2007.03.059. PMID 17659962